CLINICAL TRIAL: NCT06043986
Title: Would Artifical Intelligence Reduce Delays to Nurse Response Times
Brief Title: Would Artificial Intelligence Reduce Delays to Nurse Response Times
Acronym: WAiRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CD22/153868
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Nurse's Role

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bed bay A: Time from nurse call system activated by the novel nurse call system to initial response time T1 and time to complete task T2.
  Reason for nurse call system activated: Toilet/Pain/Medication/ /Need a nurse/Other
  Interventions: Device: novel nurse call system
- Bed bay B: Time from nurse call system activated by standard system to initial response timeT1 and time to complete task T2.

INTERVENTIONS:
Device: novel nurse call system — Inavya Ventures Ltd (Inavya) has developed a medical-grade artificial intelligence enabled mobile system (AVATR) to support out-of-hospital healthcare. AVATR is approved as a UK Government official supplier of healthcare technology on the UK Digital Marketplace for cloud-based solutions (G Cloud). AVATR in hospital, will connect to the existing AVATR outpatient service building on existing AVATR technology, which is regulated CE-mark Grade 1 (EU/UK). The research team will create, deploy and test a novel ward-based AI technology innovation to transform current nurse call systems to patient-centred mobile technology assets at bedside, thus reducing the need for unproductive visits by nurses to the bedside, which takes away time and attention where it is otherwise best served.
  Having mobile connection to the patients, would improve patient experience and saving nursing staff time, thereby improving quality of care, and saving money.
  Groups: Bed bay A

SUMMARY:
Patients are admitted to wards at all times of day and night and in various states of ill health. As this research is non interventional and does not impact on patient safety, the guidance from the ethics committee was reviewed and agreed that it would be appropriate to enrol every admission into the 2 bed bays and gain consent within 24 hours of admission.All data collected within the trial using the smart tablets will be associated to a study number, no patient details will be stored on the smart tablet and therefore the cloud data store.It has been discussed with the trust information governance and this complies with their regulations.

Any patient identifiable data will be kept by the research team. All data will be archived and stored as per the Sponsors policy. The novel nurse call system has been designed to be user friendly to all patients regardless of age, learning ability and first language used. By using colours, images and words in the hope that this will be accessible to all. The nursing staff on the ward advised on the main reasons for the nurse call system activation and therefore the icons used in the novel system were adapted from this. This trial was discussed in the patient and public involvement group. As this is a pilot trial, any adaptions that need to be made will be made before the large scale trial.

ELIGIBILITY:
Inclusion Criteria:

All adults 18 years who are admitted to the cardiology admissions ward will be eligible to take part.

-

Exclusion Criteria: Any patient who does not wish to participate will have their anonymised data removed from the trial.

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the cardiology ward
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
study objective | 1 year
  The primary outcome of this study is the time taken to respond to the alert raised by the novel nurse call system and time taken from call to completion of task.

SECONDARY OUTCOMES:
Nursing time saved | 1 year
  The time taken using the novel system will be measured against the regular method to find the difference in time.
patient acceptability of the novel system | 1 year
  this is a qualitative measure

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No